CLINICAL TRIAL: NCT07358728
Title: OSIA System Bilateral Implantation Efficacy Evaluation in Children With Ear Aplasia
Acronym: APLOSIA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP250940; IDRCB (Other: 2025-A01943-46)
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Deafness Caused by High Grade Microtia or Ear Atresia
Keywords: Microtia; Ear atresia; Deafness; Surgery; Hearing aid; Hearing implant
MeSH Terms: conditions — Congenital Microtia; Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral OSIA2 Implantation (Experimental): Bilateral implantation of two OSIA2 implants during a standard care surgery.
  Interventions: Other: Audiological tests; Behavioral: Speech, Spatial and Qualities of Hearing Scale

INTERVENTIONS:
Other: Audiological tests — FraSIMAT (French Simplified Matrix Test) and ERKI tests will be performed with one activated implant versus both activated 6 months after surgery
Behavioral: Speech, Spatial and Qualities of Hearing Scale — The patients will answer the SSQ (Speech, Spatial and Qualities of Hearing Scale) 6 months after his surgery.

SUMMARY:
The aim of this study is to compare speech perception in noise with one activated Osia (unilateral) versus two activated Osia (bilateral), in children with high grade microtia/ear atresia fitted with bilateral Osia implants. In order to do these measurements, the enrolled children will get OSIA implants on both sides during a standard surgery procedure. Six months following the implantation, audiologist testing will be done with one implant active compared to both.

DETAILED DESCRIPTION:
High grade microtia corresponds to a congenital malformation of the pinna and the external auditory meatus associated with a malformation of the middle ear. Ear atresia a congenital malformation of the external auditory meatus and middle ear, associated to a normal or near norma pinna.

In the case of hearing loss related to high grade microtia or ear atresia, be the type of hearing rehabilitation cannot be achieved with conventional air-conduction hearing aids, due to the absence of an ear canal. Different options are available and reimbursed by French medical insurance system. The Cochlear Osia implant is a semi-implantable bone conduction hearing aids. It is an active, transcutaneous (closed-skin) implant, which has the CE mark and is covered by the Health Insurance Fund for adults.

When deafness is bilateral and unaided, it impacts the development of oral language, daily life, and academic progress. Studies also show that speech perception in noisy environments is impaired. This can be very disabling, especially for young school-aged children. There are also studies showing that sound localization is improved when using two hearing aids.

Although bilateral fitting has benefits, bone conduction hearing aids are not always surgically placed bilaterally in children with ear aplasia and no clinical research has yet been conducted with the OSIA system. The objective of this study is to evaluate the effectiveness of bilateral implantation of the Osia System in children with high grade microtia or ear atresia.

Once the implantation surgery is done, the patient will come back for at least three visits: two adjustment visits, 1 month and 5 months afterwards, and two ENT consultations at 1 month and 6 months. These visits are part of the usual follow-up for children with bone conduction implants. Experimental audiological measurements will be carried out at the 6-month visit.

ELIGIBILITY:
Inclusion Criteria:

* To be aged between 7 and 17 years old at the time of enrolment
* Use spoken French as primary mode of communication
* Diagnostic of moderate to severe bilateral high grade microtia and/or ear atresia resulting in conductive hearing loss with an ACPTA between 60 and 80 dB and a BCPTA between 0 and 20 dB
* Fitted with a unilateral or bilateral headband/headband/adhesive bone conduction device for more than 12 months.
* In case of microtia: after or before ear reconstruction planned using the conventional costal cartilage graft procedure; anatomical conditions allowing implantation of the OSIA outside the area of a future ear reconstruction.
* To be a medical and audiological candidate for the OSIA system
* To be affiliated with a health insurance plan or be eligible for it
* Signed consent from the legal guardian(s)

Exclusion Criteria:

* Weight less than 7 kg (CE marking limit)
* Diagnosed with a severe neurological condition, identified by an MRI and/or a neuropediatric assessment
* Diagnosed with a severe cognitive impairment, child psychiatric impairment, or developmental delay
* Diagnosed with a severe cochleovestibular or cochlear nerve malformation
* Live in a social context that does not allow for long-term follow-up
* To be part of a family that does not understand spoken French
* Already equipped with one (or two) bone conduction implant(s)
* Affiliated with minimum state healthcare (AME)
* To currently be pregnant or breastfeeding

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Implantation success | 6 months
  Successful bilateral versus unilateral implantation identified as an increase of at least 3 dB RSB (signal-to-noise ratio) with bilateral conditions compared to unilateral condition value.

SECONDARY OUTCOMES:
Prosthetic gain | 5 months
  Prosthetic gain measured by preoperative pure-tone and speech audiometry with the removable device preoperatively and with ipsilateral OSIA:
Prosthetic gain | 6 months
  - Prosthetic gain in pure-tone audiometry (difference in mean air conduction with and without the device)
Prosthetic gain | 6 months
  - Prosthetic gain in speech audiometry (difference in SRT (Speech Reception Threshold) with and without the device)
Security and skin tolerance | 6 months
  Occurrence of adverse events/serious adverse events, particularly skin complications (hematoma, local injection, skin erosion related to magnetization)
Sound localization | 6 months
  ERKI localization test with one activated OSIA versus two activated OSIAs
Hearing quality | 6 months
  Speech and spatial hearing quality scale using the SSQ questionnaire (Speech, Spatial and Qualities of Hearing Scale) scaled between 0 (lowest quality) to 10 points (best quality)
Daily use | 6 months
  Time length use of OSIA using the data logging OSIA system

CONTACTS AND LOCATIONS:
Overall Officials: Françoise DENOYELLE, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants Malades, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No